CLINICAL TRIAL: NCT00003382
Title: A Phase I Study of Gemcitabine/Topotecan in Combination in Refractory Ovarian Cancer or Cancer of the Fallopian Tube
Brief Title: Combination Chemotherapy Consisting of Gemcitabine And Topotecan in Treating Patients With Refractory or Recurrent Ovarian or Fallopian Tube Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000066377; GOG-9702
Record Dates: First submitted 1999-11-01; First posted 2003-07-15 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2006-05

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Filgrastim; Gemcitabine; Topotecan

INTERVENTIONS:
Biological: filgrastim
Drug: gemcitabine hydrochloride
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy consisting of gemcitabine and topotecan in treating patients with refractory or recurrent ovarian or fallopian tube cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated doses of the combination of gemcitabine and topotecan administered with and without filgrastim (G-CSF) in patients with refractory ovarian or fallopian tube cancer.
* Describe and quantitate the clinical toxicities of these regimens in this patient population.

OUTLINE: This is a dose escalation study.

Patients receive gemcitabine IV over 30 minutes on days 1 and 8 and topotecan IV over 30 minutes on days 2-4. Some patients receive filgrastim (G-CSF) subcutaneously on days 9-14. Treatment repeats every 28 days for up to 5-10 courses.

Cohorts of 3-6 patients receive escalating doses of topotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose below that at which 2 of 6 patients experience dose limiting toxicity (DLT). Dose escalation of gemcitabine then continues in cohorts of 3-6 patients until the MTD is determined. The MTD is defined as the dose below that at which 2 of 6 patients experience DLT.

Patients are followed every 2-3 months for 2 years, every 6 months for 3 years, then annually thereafter.

PROJECTED ACCRUAL: Approximately 24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically documented refractory or recurrent ovarian epithelial or fallopian tube cancer
* No borderline ovarian cancer
* Extra-ovarian papillary serous tumors eligible
* Must not be eligible for any higher priority phase II or III GOG protocol

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* GOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* SGOT no greater than 3 times upper limit of normal (ULN)
* Bilirubin no greater than 1.5 mg/dL
* Elevated levels of alkaline phosphatase allowed

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No angina pectoris or clinically significant multifocal uncontrolled cardiac dysrhythmias
* No uncontrolled hypertension

Other:

* No other active malignancy
* No prior malignancy within the past 5 years except nonmelanomatous skin cancer
* No active infection
* No underlying medical problem that would prevent compliance
* No known hypersensitivity to E. coli-derived drug preparations
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Must have received at least 1 prior platinum- and paclitaxel-based regimen
* At least 4 weeks since prior chemotherapy
* No prior topotecan and/or gemcitabine
* No prior chemotherapy for a different prior malignancy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to more than 10% of bone marrow
* At least 2 weeks since limited field radiation therapy

Surgery:

* Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-05; Primary Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ming-teh D. Chen, MD, Study Chair — Women's Cancer Center - Los Gatos
Locations (6):
- United States (6):
  - Community Hospital of Los Gatos, Los Gatos, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Women's Cancer Center, Palo Alto, California
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Chen MD, Fleming GF, Mitchell S, Horowitz I. A phase I trial of gemcitabine and topotecan in previously treated ovarian or peritoneal cancer: a Gynecologic Oncology Group study. Gynecol Oncol. 2006 Jan;100(1):111-5. doi: 10.1016/j.ygyno.2005.07.114. Epub 2005 Sep 8. PMID 16150481